CLINICAL TRIAL: NCT04130191
Title: A Three-year, Non-interventional, Prospective, Multicenter Study to Evaluate the Long- Term Effectiveness of Lanadelumab in Real-world Clinical Practice (ENABLE)
Brief Title: A Study of Lanadelumab in Persons With Hereditary Angioedema (HAE) Type I or II
Acronym: ENABLE
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP643-402; TAK-743-402 (Other: Takeda Development Center Americas)
Record Dates: First submitted 2019-10-03; First posted 2019-10-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with hereditary angioedema (HAE): Participants who initiate treatment with lanadelumab according to current product labelling will be enrolled and followed for up to 24 or 36 months (depending on their enrollment date).

SUMMARY:
The main aim of this study is to compare the number of HAE attacks occuring in persons using lanadelumab with the number of HAE attacks before lanadelumab treatment was started.

Data from participants who start the study after 1 March 2021, will be collected for 24 months; data from all other participants (who started the study before 1 March 2021) will be collected for 36 months. Participants will report information in a smartphone application at study start and for the next 3 months and then every 6 months until the study ends; data will also be collected by the study doctor during routine clinic visits

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provision of written, signed, and dated (personally or via a legally authorized representative) informed consent to participate in the study.
* Initiation of treatment with lanadelumab in accordance with current product labelling. Decision to start treatment with lanadelumab must be made before and be independent from enrollment in the study.
* Availability of information for HAE attack-related variables assessed at study enrollment for the previous three months.
* Ability to use a smartphone for data collection in this study.

Exclusion Criteria:

* Inability to provide written, signed, and dated informed consent.
* Participation in the study not considered appropriate by the treating physician/investigator.
* Contraindication to treatment with lanadelumab according to current product labelling.
* Pregnant or breastfeeding.
* Concomitant exposure to any investigational therapy (including medications not used for HAE).
* Current or planned participation in other interventional studies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with type 1 or type 2 HAE who initiate treatment with lanadelumab according to the current product labelling.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Incidence Rate Ratio of On-Treatment Participant-Reported Hereditary Angioedema (HAE) Attacks | Up to 36 months
  HAE attack is defined as a discrete episode during which the participant progress from no angioedema to symptoms of angioedema. Incidence rate ratio of on-treatment patient-reported HAE attacks up to three years after initiation of lanadelumab compared to the history of HAE attacks of last three months prior to lanadelumab use will be reported.

SECONDARY OUTCOMES:
Rate of On-Treatment Participant-Reported Hereditary Angioedema (HAE) Attacks From Day 70 | From Day 70 up to 36 months
  Rate of participant-reported HAE attacks during treatment with lanadelumab from day 70 will be assessed.
Rate of Mild, Moderate, Severe Hereditary Angioedema (HAE) Attacks | Up to 36 months
  The overall severity of attack is determined using following definitions: mild (Temporary or mild discomfort), moderate (Activity limited mildly or moderately. Some assistance may be needed), severe (Activity considerably limited, assistance needed).
Number of On-Treatment Participant-Reported Hereditary Angioedema (HAE) Attacks Based on Anatomical Location | Up to 36 months
  Number of on-treatment participant-reported HAE attacks based on anatomical (peripheral, abdominal, laryngeal) location will be assessed.
Proportion of Hereditary Angioedema (HAE) Attacks for Which On-Demand Therapy is Used | Up to 36 months
  Proportion of HAE attacks for which participants use on-demand therapy will be assessed.
Time to First Hereditary Angioedema (HAE) Attack for Which On-Demand Therapy is Used | Up to 36 months
  Time to first HAE attack for which on-demand therapy is used will be assessed.
Proportion of Hereditary Angioedema (HAE) Attacks Requiring Visit to an Healthcare Provider (HCP), Access to an Emergency Room (ER), or Hospitalization | Up to 36 months
  Proportion of HAE Attacks requiring visit to HCP, access to an ER, or hospitalization will be assessed.
Angioedema Quality of Life (AE-QoL) | Up to 36 months
  The AE-QoL is developed to measure participant-reported health-related quality of life (HRQoL) impairment in participants with recurrent angioedema. It is a self-administered participant related outcome (PRO) with a recall period of 4 weeks. There are 17 items across 4 domains: functioning (4 items), fatigue/mood (5 items), fears/shame (6 items), and food (2 items). Responses use a 5-point Likert scale ranging from 'never' to 'very often.' Global scores range from 0 to 100 and scores by domains range from 0 to 100, where 0 indicates highest quality of life and 100 lowest quality of life.
Fatigue Severity Scale (FSS) | Up to 36 months
  Participant reported fatigue will be measured by the FSS. The FSS is a 9-item questionnaire measuring participants fatigue severity and its impact on motivation, exercise, physical functioning, and work and social life. It uses a 7-point Likert scale response (1 = strongly disagree, 7 = strongly agree) and the final score is obtained as mean of the response scores to the individual questions.
Hospital Anxiety and Depression Scale (HADS) | Up to 36 months
  The HADS is a self-rating scale developed to detect the levels of depression and anxiety experienced by participants. It is a self-administered PRO composed of 14 items, of which seven relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0 to 3, which means that a person can score between 0 and 21 for either anxiety or depression. Recommended cut-off scores are 8 to 10 for doubtful cases and greater than or equal to (> or =) 11 for definite cases.
Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9) | Up to 36 months
  The TSQM is a generic questionnaire to measure participants satisfaction with medication using yes/no and 5- or 7-point Likert scale response options. It is a self-administered PRO instrument designed for adults aged 18 years or older with a recall period of two to three weeks, or since the last medication use. Version TSQM-9 includes three domains: effectiveness (three items), convenience (three items), and global satisfaction scale (three items).
Work Productivity and Activity Impairment: General Health (WPAI:GH) | Up to 36 months
  The WPAI:GH is a generic questionnaire to measure the effect of general health and symptom severity on work productivity and regular activities during the past seven days. It can be self or interviewer-administered to adults aged 18 years or older. This six-item PRO instrument covers work (five items) and daily activities (one item) using yes/no or numerical answers (number of hours).
Adult Carer Quality of Life (AC-QoL) Questionnaire | Up to 36 months
  The AC-QoL is a 40-item tool that measures the overall QoL for adult carers, and subscale scores for eight domains of QoL: support for caring, caring choice, caring stress, money matters; personal growth; sense of value, ability to care, and carer satisfaction. It is self-administered to adult carers and should take no longer than 10 minutes to complete. Scores range from 0 to 120, with higher scores indicating greater QoL.
Dose of Lanadelumab | From start of the study up to 36 months
  Dose of lanadelumab used during the study will be assessed.
Frequency of Administration of Lanadelumab | From start of the study up to 36 months
  Frequency of lanadelumab injections during the study will be assessed.
Participants' Adherence Rate to Treatment with Lanadelumab | Up to 36 months
  Adherence is defined as the proportion of time on treatment over the study observation time period, times the proportion of actual lanadelumab doses taken per label as reported by participants through an administration diary over the total expected lanadelumab doses per label during the treatment period.
Frequency of Use of Approved Lanadelumab Dosing Regimens | Up to 36 months
  Frequency of use of approved lanadelumab dosing regimens will be assessed.
Frequency of Administration Modalities of Lanadelumab | Up to 36 months
  Frequency of administration modalities of lanadelumab (self-administration versus (vs). administration by a caregiver, HCP, or other) will be assessed.
Number of Administrations of Lanadelumab Before Participant Discontinuation | Up to 36 months
  Number of administrations of lanadelumab before participant discontinuation from the study will be assessed.
Frequency of Reasons for Discontinuation of Treatment With Lanadelumab Reported by Participants | Up to 36 months
  Frequency of reasons for discontinuation of treatment with lanadelumab reported by participants will be assessed.
Adverse Event (AE) Incidence, Type, Seriousness and Relatedness to Lanadelumab Treatment | From start of the study up to 36 months
  An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (study) product whether or not related to the medicinal product. AE incidence, type, seriousness and relatedness to lanadelumab treatment will be assessed.
Severity of Non-Serious Adverse Events (AEs) | From start of the study up to 36 months
  Severity of AEs is determined by using the following definitions: Mild: A type of AE that is usually transient and may require only minimal treatment or therapeutic intervention, the event does not generally interfere with activities of daily living. Moderate: A type of AE that is usually alleviated with specific therapeutic intervention, the event interferes with usual activities of daily living, causing discomfort, but poses no significant or permanent risk of harm to the research participant. Severe: A type of AE that interrupts usual activities of daily living (ADL), or significantly affects clinical status, or may require intensive therapeutic intervention. Severity of non-serious AEs will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (19):
- Medical University of Vienna, Vienna, Austria
- Germany (8):
  - Klinikum der Johann-Wolfgang Goethe-Universitat, Frankfurt am Main, Hesse
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Universitatsklinikum Schleswig-Holstein, Lübeck
  - Hämophilie Zentrum Rhein Main GmbH, Mörfelden-Walldorf
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Ulm, Ulm
- Israel (2):
  - Bnai Zion Medical Center, Haifa
  - Sheba Medical Center - PPDS, Ramat Gan
- Italy (3):
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - ASST Fatebenefratelli Sacco - Ospedale Luigi Sacco, Milan
  - Azienda Ospedale Università Padova, Padua
- Al-Rashed Allergy Center, Kuwait City, Kuwait
- Spain (2):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Luzerner Kantonsspital LUKS, Lucerne

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment? commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Zanichelli A, Wuillemin WA, Aygoren-Pursun E, Banerji A, Busse PJ, Betschel SD, Cancian M, Gagnon R, Goodyear MD, Kinaciyan T, Kessel A, Magerl M, Recke A, Wedner HJ, Estepan DN, Watt M, Andresen I, Juethner S, Khutoryansky N, Martinez-Saguer I. Lanadelumab's impact on hereditary angioedema control and quality of life across disease activity subgroups: Real-world evidence. Ann Allergy Asthma Immunol. 2025 Nov;135(5):560-569.e2. doi: 10.1016/j.anai.2025.07.025. Epub 2025 Sep 6. PMID 40769455
- [Derived] Tachdjian R, Banerji A, Busse PJ, Agmon-Levin N, Anderson J, Cancian M, Spadaro G, Enciu C, Estepan DN, Khutoryansky N, Jain S, Recke A. Effective long-term prophylaxis with lanadelumab in adolescents with hereditary angioedema: EMPOWER/ENABLE. Pediatr Allergy Immunol. 2025 Apr;36(4):e70072. doi: 10.1111/pai.70072. PMID 40171989
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fdc4db2bf003ab47313